CLINICAL TRIAL: NCT00072618
Title: A Phase I/II Multi-Center Study of Weekly Taxotere (Docetaxel) in Combination With Aptosyn (Exisulind) in Non-Small Cell Lung Cancer (NSCLC) Patients Who Have Failed a Prior Platinum-Containing Regimen
Brief Title: Phase II Study of Taxotere in Combination With Exisulind in Non-Small Cell Lung Cancer (NSCLC) Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 026B; NCT00036010 (obsolete NCT alias)
Record Dates: First submitted 2003-11-05; First posted 2003-11-07 (Estimated); Last update posted 2011-10-20 (Estimated); Status verified 2011-10

CONDITIONS: NSCLC
MeSH Terms: interventions — sulindac sulfone

INTERVENTIONS:
Drug: Exisulind

SUMMARY:
The purpose of this study is to determine if the combination of Taxotere and exisulind is an effective and safe treatment for patients with advanced NSCLC who have failed a prior platinum-containing regimen.

ELIGIBILITY:
Inclusion Criteria:

Histologically documented advanced cancer or advanced platinum-refractory non-small cell lung cancer. Platinum refractory defined as progressive disease during a platinum regimen or within 6 months following treatment.

Negative serum pregnancy test, if fertile female. Have not taken sulindac (Clinoril®) on regular basis for any indication for one week prior to enrollment and willing to remain off of sulindac for the duration of the study.

> 18 years or of legal age. Male patients, or non-pregnant and non-lactating female patients either using adequate birth control (oral contraceptives or Provera), surgically sterile or post-menopausal.

Willingness to remain off chronic NSAIDs (with the exception of ibuprofen, naproxen, or aspirin) for duration of the study. Low dose aspirin for cardiovascular prevention is acceptable.

No treatment with any other chemotherapy or radiotherapy within 2 weeks prior to entering the study.

Exclusion Criteria:

Any condition or any medication which may interfere with the conduct of the study.

Known hypersensitivity to sulindac (Clinoril®) or taxanes. Use of an investigational medication or device within one month of initiating study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52
Dates: Start 2001-10; Study Completion 2003-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Colorado Health Sciences Center, Aurora, Colorado
  - University of Chicago Medical Center, Chicago, Illinois